CLINICAL TRIAL: NCT02944214
Title: Compare the Renal Protective Effects of Febuxostat and Benzbromarone in Middle-to-late Stages of Chronic Kidney Disease Patients: a Multi-center Randomized Controlled Study
Brief Title: Compare the Renal Protective Effects of Febuxostat and Benzbromarone in CKD Chinese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ai Peng, Professor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FB2016MC
Record Dates: First submitted 2016-10-20; First posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Kidney Disease; Hyperuricemia; Abnormal Renal Function
Keywords: Hyperuricemia; Renal Function; Chronic kidney disease; Febuxostat; Benzbromarone
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperuricemia | interventions — Febuxostat; Benzbromarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Febuxostat (Experimental): take orally,10-80mg per day, for 1 year,start with a low dose, and adjust the dose according to the level of uric acid
  Interventions: Drug: Febuxostat
- Benzbromarone (Experimental): take orally,12.5-100mg per day, for 1 year,start with a low dose, and adjust the dose according to the level of uric acid
  Interventions: Drug: Benzbromarone

INTERVENTIONS:
Drug: Febuxostat — It acts as an inhibitor of xanthine oxidase, thus lowering urate concentrations in the body
  Other Names: Uloric; Adenuric
  Arms: Febuxostat
Drug: Benzbromarone — It is structurally related to the antiarrhythmic amiodarone, and it is a uricosuric agent and non-competitive inhibitor of xanthine oxidase
  Other Names: Desuric
  Arms: Benzbromarone

SUMMARY:
The purpose of this study is to determine whether febuxostat and benzbromarone could protect renal function in chinese, and which one could be better.

DETAILED DESCRIPTION:
Chronic kidney disease patients with hyperuricemia and glomerular filtration rate (GFR) 20-60 ml/min were treated by febuxostat or benzbromarone. Follow up the changes of serum uric acid, serum creatinine and GFR levels. Compare the effects on renal function of these two drugs.

ELIGIBILITY:
Inclusion Criteria:

Chronic kidney disease patients with glomerular filtration rate (GFR,20-60ml/min) who match one of the following criteria:

1. Gout
2. serum uric acid > 480umol/L

Exclusion Criteria:

1. GFR<20ml/min or GFR >60ml/min
2. Liver dysfunction (Aspartate transaminase or/and alanine aminotransferase exceed 2 times of normal range)
3. Urinary tract obstruction
4. unstable angina, heart failure (stage III-IV, NYHA), new stroke, need diuretics for long-term treatment
5. Severe lung diseases or cancers
6. Pregnant woman or woman who prepare to be pregnant，nursing mothers
7. unable to sign informed consent form，or disagree with following-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
serum creatinine, estimated glomerular filtration rate (eGFR) | up to 12th months
  eGFR will be estimated by CKD-EPI equation, which is most widely used recently in the world. eGFR will be calculated according to serum creatinine, age, gender and race.

SECONDARY OUTCOMES:
urine protein | 6th months, 12th months
adverse drug reaction | 1st month, 2nd months, 3rd months, 6th months, 9th months, 12th months

CONTACTS AND LOCATIONS:
Overall Officials: Ai Peng, MD, PhD, Study Chair — Department of Nephrology & Rheumatology, Shanghai Tenth People's Hospital
Locations (1):
- Department of Nephrology & Rheumatology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No